CLINICAL TRIAL: NCT03501602
Title: Comparison of Endotracheal Intubation Over the Aintree Catheter With Fiberoptic Bronchoskop Via the I-gel and Laryngeal Mask Airway Protector
Brief Title: Comparison of Endotracheal Intubation Over the Aintree With Fiberoptic Bronchoskop Via the I-gel and LMA Protector
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Aslı duygu aydaş, specialist doctor, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/77
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Intubation;Difficult
Keywords: aintree, LMA protector; I-gel LMA, Fiberoptic Bronchoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LMA protector group (Active Comparator): The LMA Protector is a single use supraglottic airway device. This airway device provides access and functional separation of the respiratory and digestive tracts
  Interventions: Device: LMA protector
- I-gel LMA group (Active Comparator): The I-gel is an alternative supraglottic device which provides the seal over the airway versus an inflatable cuff.
  Interventions: Device: I-gel LMA

INTERVENTIONS:
Device: LMA protector — In this arm the LMA protector will be inserted. The time from took the LMA to placement of the LMA will be recorded. In patients with adequate ventilation, an Aintree catheter placed on a fiberoptic bronchoscope in LMA will be delivered. Cord vocals will be seen on the monitor and the aintree catheter will be sent into the trachea. After the insertion of the trachea, the fiberoptic bronchoscope and LMA are removed and the patient's intubation tube is advanced through the Aintree catheter to the patient's trachea. Once you have made sure that the tube is in the trachea, it will be removed. The time from insertion of the LMA to placement of the endotracheal tube will be recorded.
  Other Names: aintree catheter, Fiberoptic brochoscop
  Arms: LMA protector group
Device: I-gel LMA — In this arm the I-gel LMA will be inserted. The time from took the LMA to placement of the LMA will be recorded. In patients with adequate ventilation, an Aintree catheter placed on a fiberoptic bronchoscope in LMA will be delivered. Cord vocals will be seen on the monitor and the aintree catheter will be sent into the trachea. After the insertion of the trachea, the fiberoptic bronchoscope and LMA are removed and the patient's intubation tube is advanced through the Aintree catheter to the patient's trachea. Once you have made sure that the tube is in the trachea, it will be removed. The time from insertion of the LMA to placement of the endotracheal tube will be recorded.
  Other Names: aintree catheter, Fiberoptic brochoscop
  Arms: I-gel LMA group

SUMMARY:
Investigators aimed to compare the ease of use of the LMA protector and I-gel LMA for tracheal intubation with the Aintree catheter in our study.

Laryngeal mask airway (LMA) protector is the second generation perilaryngeal seal type supraglottic airway tool. The I-gel LMA is the second generation uncuffed supraglottic airway device. The Aintree Intubation Catheter has been designed for assisted fiberoptic intubation and for uncomplicated, atraumatic endotracheal tube exchange.Both LMA types have a structure that permits endotracheal intubation. In cases of difficult intubation, these two LMA types can be used. In the literature, there is no study comparing these two LMA types using Aintree catheter.Difficult Airway Society (DAS) published a guide for tracheal intubation in 2011 using Aintree. According to this guide, LMA type LMA Supreme is the most unfavorable for this process. However, there is no research or recommendation on the type of LMA most suitable for use in the literature. In accordance with the data of this study, it will be tried to show which LMA type may be suitable for intubation with Aintree catheter in patients.

DETAILED DESCRIPTION:
Investigators will include adult patients over 18 years of age who will undergo a surgical operation requiring intubation. Patients will be divided into protector LMA and I-gel LMA groups by closed envelope method. Forty patients are planned for both groups. The age, weight, height, body mass index (BMI) of the patients, operation to be performed, ASA, mallampati, thyromental distance values will be recorded. A standard induction of anesthesia will be applied to the patient. After 2 minutes the LMA will be inserted. It will be recorded how many numbered LMAs are used, success rate, number of trials, optimization maneuver required. With LMA, whether sufficient amount of tidal volume can be given to the patient and whether sufficient amount of chest departure is observed during ventilation will be recorded together with tidal volume values. In patients with adequate ventilation, an Aintree catheter placed on a fiberoptic bronchoscope in LMA will be delivered. Fiberoptic laryngeal appearance staging will be performed:

Stage 4: only the cords look Stage 3: cords + posterior epiglot seen Stage 2: cords + anterior epiglot seen Stage 1: no cords seen Cord vocals will be seen on the monitor and the aintree catheter will be sent into the trachea. After insertion of the trachea, the fiberoptic bronchoscope and LMA are removed and the patient's intubation tube is advanced through the Aintree catheter in the appropriate size and the tube is placed in the trachea. Once participants have made sure that the tube is trachea, it will be removed. The time from insertion of the LMA to placement of the endotracheal tube will be coded. During the procedure, the patient's blood pressure, heart rate, oxygen saturation, any complications that may develop will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Be intubated in surgical operation requiring intubation
* over 18 years old

Exclusion Criteria:

* Difficult intubation story
* Difficult intubation risk
* Presence of gastric reflux

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-04-05 (Estimated); Study Completion 2019-07-05 (Estimated)

PRIMARY OUTCOMES:
Time to Successful Tracheal Intubation | Up to 10 minutes
  This measure of time begins with the handling of the supraglottic device to confirming the appropriate placement of the device by noting the presences of end tidal carbon dioxide.

SECONDARY OUTCOMES:
Time to Placement of the Supra Glottic Device | Up to 10 minutes
  This measure of time begins with the handling of the supra glottic device to confirming the appropriate placement of the device by noting the presences of end tidal carbon dioxide
Time to Placement of the Aintree Airway Intubation Catheter | Up to 10 minutes
  This measure of time begins with the handling of the fiberscope to withdrawal of the fiberscope from the Aintree and setting the fiberscope down
Laryngeal appearance staging | Up to 10 minutes
  Stage 4: only the cords look Stage 3: cords + posterior epiglot seen Stage 2: cords + anterior epiglot seen Stage 1: no cords seen

OTHER OUTCOMES:
Mouth openness | Up to 10 minutes
  measuring the maximum openness the patient can open his mouth
thiromental distance | Up to 10 minutes
  The distance between the lowest end of the jaw and the thyroid overhang when the head is in full extension.
pre-induction systolic and diastolic pulse | Up to 10 minutes
  pre-induction systolic and diastolic pulse rate measurement
pre-induction heart rate | Up to 10 minutes
  pre-induction heart rate measurement
pre-induction oxygen saturation | Up to 10 minutes
  pre-induction oxygen saturation measurement
systolic and diastolic pulse after LMA insertion | Up to 10 minutes
  systolic and diastolic pulse rate measurement after LMA insertion
heart rate after LMA insertion | Up to 10 minutes
  heart rate measurement after LMA insertion
oxygen saturation after LMA insertion | Up to 10 minutes
  oxygen saturation measurement after LMA insertion
systolic and diastolic pulse after intubation | Up to 10 minutes
  systolic and diastolic pulse rate measurement after intubation
heart rate after after intubation | Up to 10 minutes
  heart rate measurement after intubation
oxygen saturation after intubation | Up to 10 minutes
  oxygen saturation measurement after intubation
end tidal carbon dioxide after LMA insertion | Up to 10 minutes
  end tidal carbon dioxide measurement after LMA insertion
end tidal carbon dioxide after intubation | Up to 10 minutes
  end tidal carbon dioxide measurement after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Kemal T Saraçoğlu, assoc. prof., Study Chair — Sağlık Bilimleri Üniversitesi Kocaeli Derince Eğitim ve Araştırma Hastanesi
Locations (1):
- Aslı Duygu Aydaş, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided